CLINICAL TRIAL: NCT05168813
Title: Multi-Center, Randomized, Efficacy Study of COVID-19 mRNA Vaccine in Regions With SARS-CoV-2 Variants of Concern
Brief Title: Efficacy Study of COVID-19 mRNA Vaccine in Regions With SARS-CoV-2 Variants of Concern
Acronym: CoVPN3008
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: COVID-19 Prevention Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CoVPN 3008; UM1AI068614 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2021-12-23 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2 Infection; HIV Infections; COVID-19
Keywords: SARS-CoV-2; HIV; COVID-19
MeSH Terms: conditions — COVID-19; HIV Infections | interventions — 2019-nCoV Vaccine mRNA-1273; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Study Group 1 (Experimental): COVID-19 mRNA vaccine in 100 mcg dose to be administered as an IM injection into the deltoid muscle on Months 0, 1, and 6 among adults living with HIV who are SARS-CoV-2 negative at baseline.
  Interventions: Biological: Moderna mRNA-1273; Biological: Moderna mRNA-1273.222; Biological: Vaccine 3 Dose
- Study Group 2 (Experimental): COVID-19 mRNA vaccine in 100 mcg dose to be administered as an IM injection into the deltoid muscle on Months 0 and 6 among adults living with HIV who are SARS-CoV-2 positive at baseline.
  Interventions: Biological: Moderna mRNA-1273; Biological: Moderna mRNA-1273.222; Biological: Vaccine 2 Dose
- Study Group 3 (Experimental): COVID-19 mRNA vaccine in 100 mcg dose to be administered as an IM injection into the deltoid muscle on Months 0, 1, and 6 among HIV negative adults who are SARS-CoV-2 negative at baseline.
  Interventions: Biological: Moderna mRNA-1273; Biological: Moderna mRNA-1273.222; Biological: Vaccine 3 Dose
- Study Group 4 (Experimental): COVID-19 mRNA vaccine in 100 mcg dose to be administered as an IM injection into the deltoid muscle on Months 0 and 6 among HIV negative adults who are SARS-CoV-2 positive at baseline.
  Interventions: Biological: Moderna mRNA-1273; Biological: Moderna mRNA-1273.222; Biological: Vaccine 2 Dose
- Monovalent (Experimental): mRNA-1273 vaccine in 100 mcg dose to be administered as an IM injection into the deltoid muscle on Month 6.
  Interventions: Biological: Moderna mRNA-1273
- Bivalent (Experimental): mRNA-1273.222 vaccine in 100 mcg dose to be administered as an IM injection into the deltoid muscle on Month 6.
  Interventions: Biological: Moderna mRNA-1273.222

INTERVENTIONS:
Biological: Moderna mRNA-1273 — COVID-19 vaccine (mRNA-1273) developed by Moderna, Inc. is a lipid nanoparticle (LNP) dispersion of a messenger ribonucleic acid (mRNA) encoding the prefusion stabilized S protein of SARS-CoV-2 formulated in LNPs composed of 4 lipids (1 proprietary and 3 commercially available).
  Arms: Monovalent; Study Group 1; Study Group 2; Study Group 3; Study Group 4
Biological: Moderna mRNA-1273.222 — COVID-19 vaccine (mRNA-1273.222) developed by Moderna, Inc. is an updated bivalent version of Moderna's mRNA-1273 vaccine, composed of equal parts of mRNA-1273 and mRNA that encodes the S protein of the Omicron subvariants BA.4/.5 (which have the same S protein).
  Arms: Bivalent; Study Group 1; Study Group 2; Study Group 3; Study Group 4
Biological: Vaccine 3 Dose — COVID-19 mRNA vaccine in 100 mcg dose given as IM injection into the deltoid muscle on Months 0, 1, and 6.
  Arms: Study Group 1; Study Group 3
Biological: Vaccine 2 Dose — COVID-19 mRNA vaccine is to be administered as IM injection into the deltoid muscle on Months 0 and 6.
  Arms: Study Group 2; Study Group 4

SUMMARY:
The study will evaluate the clinical efficacy of different dosing regimens of the Moderna COVID-19 mRNA vaccine (100 mcg) in preventing COVID-19 disease in people who are living with HIV or have comorbidities associated with elevated risk of severe COVID-19, with the different vaccine regimens assessed determined by whether the participant had evidence of prior SARS-CoV-2 infection at enrollment.

DETAILED DESCRIPTION:
The study is constructed to help inform which vaccine regimen, likely in combination with enhanced HIV care, could serve as a public health model for an effective and cost-efficient approach to preventing SARS-CoV-2 disease, prolonged viral shedding, and the emergence of VOCs within this population. Moreover, we will evaluate whether immune responses postvaccination can be correlated to these clinically important outcomes.

The study will enroll 15,600 adults from many clinics in Eastern and Southern Africa. All participants in the study will get the study vaccine. There are 4 primary groups in this study. The groups differ in the number of doses of the study vaccine administered. The groups are organized by whether or not people are living with HIV and whether or not people have evidence of prior SARS-CoV-2 infection in their blood.

Group 1 includes people living with HIV and Group 3 includes people who are not living with HIV. All people in groups 1 and 3 will have no evidence of prior SARS-CoV-2 infection in their blood. Participants in Group 1 or Group 3 will get three doses of the study vaccine.

Group 2 includes people living with HIV and Group 4 includes people who are not living with HIV. All people in groups 2 and 4 will have evidence of prior SARS-CoV-2 infection in their blood. Participants in Group 2 or Group 4 will get two doses of the study vaccine.

There are 8 scheduled clinic visits over 18 months. Study visits may include physical examinations, medical history, vaccine injections, HIV testing, blood collection, nasal swabs, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

1. Age ≥ 18 years if participant self-reports living with HIV or another comorbidity known to be associated with severe COVID-19, for example (CDC.gov for exhaustive list):

   * Hypertension
   * Type 2 diabetes mellitus
   * Overweight, obese, or severely obese (ie, body mass index [BMI] ≥ 25 kg/m2)
   * Heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
   * Chronic kidney disease
   * COPD (chronic obstructive pulmonary disease)
   * Cancer
   * Non-HIV immunocompromised state (weakened immune system) or solid organ transplant
   * Pregnancy
   * Sickle cell disease
   * Smoking
2. Willingness to be followed and remain in the catchment area for the planned duration of the study.
3. Ability and willingness to provide informed consent.
4. Willingness to discuss HIV infection status, undergo related testing/monitoring labs, and receive counseling and referrals to minimize HIV acquisition/improve HIV care as appropriate based on their infection status.
5. Assessment of Understanding (AoU): Participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination with demonstration of understanding of all questionnaire items answered incorrectly.
6. Agrees not to enroll in another interventional study of an investigational research agent until after the study is completed and all the data has been obtained. Enrollment in studies of investigational research agents for the treatment of COVID-19 is allowed for participants who develop COVID-19 disease.

Exclusion Criteria:

General

1. Acutely ill 72 hours prior to or at screening. Participants meeting this criterion may be rescheduled within the relevant window periods. Participants with minor illnesses can be enrolled at the discretion of the investigator.
2. History of angioedema or anaphylaxis.

   Vaccines and other injections
3. Prior receipt of a SARS-CoV-2 vaccine.
4. History of severe allergic reaction to any ingredient of this vaccine (lipids (SM-102, polyethylene glycol [PEG] 2000 dimyristoyl glycerol [DMG], cholesterol, and 1,2-distearoyl-sn-glycero-3-phosphocholine [DSPC]), tromethamine, tromethamine hydrochloride, acetic acid, sodium acetate trihydrate, and sucrose).
5. Live attenuated vaccines received within 30 days before first vaccination (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine, live attenuated zoster vaccine).
6. Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, human papilloma virus (HPV), pneumococcal, Hepatitis A or B).
7. Blood products, systemic immunoglobulins, or monoclonal antibodies (including against SARS-CoV-2) received within 90 days before first vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14237 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Garrett, Study Chair — Centre for the AIDS Programme of Research in South Africa (CAPRISA); Philip Kotze, Study Chair — Qhakaza Mbokodo Research Clinic; Sufia Dadabhai, Study Chair — Blantyre CRS / Johns Hopkins Research Project; Nyaradzo Mgodi, Study Chair — University of Zimbabwe Clinical Trials Research Centre
Locations (47):
- Gaborone CRS, Gaborone, Botswana
- Eswatini Prevention Center CRS, Mbabane, Hhohho Region, Eswatini
- Kenya (3):
  - Moi University Clinical Research Centre, Eldoret
  - Kisumu - Kombewa CRS, Kisumu
  - Kisumu Crs, Kisumu
- Malawi (2):
  - Blantyre CRS, Blantyre
  - Malawi CRS, Lilongwe
- South Africa (32):
  - Synergy Biomed Research Institute, East London, Eastern Cape
  - Nelson Mandela Academic Research Unit CRS, Mthatha, Eastern Cape
  - PHOENIX Pharma (Pty) Ltd, Port Elizabeth, Eastern Cape
  - Josha Resarch CRS, Bloemfontein, Free State
  - MeCRU CRS, Ga-Rankuwa, Gauteng
  - Clinical HIV Research Unit (CHRU)/ Helen Joseph CRS, Johannesburg, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - Soweto - Bara CRS, Johannesburg, Gauteng
  - Wits RHI Ward 21 CRS, Johannesburg, Gauteng
  - MERC Kempton Park, Pretoria, Gauteng
  - Synexus Stanza Clinical Research Centre (CRS), Pretoria, Gauteng
  - Tembisa Clinic 4 CoVPN CRS, Tembisa, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Tongaat CRS, Durban, KwaZulu-Natal
  - Vulindlela CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Isipingo, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic CRS, Ladysmith, KwaZulu-Natal
  - MERC Middelburg, Middelburg, Mpumalanga
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
  - Rustenburg CRS, Rustenburg, North West
  - Emavundleni CRS, Cape Town, Western Cape
  - FAM-CRU (Family Clinical Research Unit), Cape Town, Western Cape
  - Groote Schuur HIV CRS, Cape Town, Western Cape
  - Masiphumelele Clinical Research Site (MASI) CRS, Cape Town, Western Cape
  - TASK Central, Cape Town, Western Cape
  - Univeristy of Cape Town Lung CRS Institute, Cape Town, Western Cape
  - TASK Eden, George, Western Cape
  - Synexus Helderberg, Stellenbosch, Western Cape
  - Ndlovu Research Centre CoVPN CRS, Elandsdoorn
  - Kliptown Soweto CRS, Johannesburg
  - PHRU Matlosana CRS, Klerksdorp
  - MERC Welkom, Welkom
- Uganda (4):
  - UVRI-IAVI HIV Vaccine Program LTD. CRS, Entebbe
  - Baylor-Uganda CRS, Kampala
  - Joint Clinical Research Centre, Kampala
  - MU-JHU Research Collaboration CRS, Kampala
- Zambia (4):
  - Cfhrz Crs, Lusaka
  - Matero Reference Clinic CRS, Lusaka
  - UNC Global Projects / Kamwala District Health Centre, Lusaka
  - Zambia Emory HIV Research Project - Ndola CoVPN CRS, Ndola

REFERENCES:
- [Result] Garrett N, Tapley A, Hudson A, Dadabhai S, Zhang B, Mgodi NM, Andriesen J, Takalani A, Fisher LH, Kee JJ, Magaret CA, Villaran M, Hural J, Andersen-Nissen E, Ferarri G, Miner MD, Le Roux B, Wilkinson E, Lessells R, de Oliveira T, Odhiambo J, Shah P, Polakowski L, Yacovone M, Samandari T, Chirenje Z, Elyanu PJ, Makhema J, Kamuti E, Nuwagaba-Biribonwoha H, Badal-Faesen S, Brumskine W, Coetzer S, Dawson R, Delany-Moretlwe S, Diacon AH, Fry S, Gill KM, Ebrahim Hoosain ZA, Hosseinipour MC, Inambao M, Innes C, Innes S, Kalonji D, Kasaro M, Kassim P, Kayange N, Kilembe W, Laher F, Malahleha M, Maluleke VL, Mboya G, McHarry K, Mitha E, Mngadi K, Mda P, Moloantoa T, Mutuluuza CK, Naicker N, Naicker V, Nana A, Nanvubya A, Nchabeleng M, Otieno W, Potgieter EL, Potloane D, Punt Z, Said J, Singh Y, Tayob MS, Vahed Y, Wabwire DO, McElrath MJ, Kublin JG, Bekker LG, Gilbert PB, Corey L, Gray GE, Huang Y, Kotze P; CoVPN 3008 Ubuntu Study Team. Hybrid versus vaccine immunity of mRNA-1273 among people living with HIV in East and Southern Africa: a prospective cohort analysis from the multicentre CoVPN 3008 (Ubuntu) study. EClinicalMedicine. 2025 Jan 20;80:103054. doi: 10.1016/j.eclinm.2024.103054. eCollection 2025 Feb. PMID 39902315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in two parts: Part A (open-label) and Part B (blinded).
Pre-assignment Details: In Part A, participants were enrolled into 4 study groups defined by baseline HIV and SARS-CoV-2 anti-S status. All ppts received mRNA-1273 at Month 0. Study groups 1 and 3 also received mRNA-1273 at Month 1. 236 ppts were excluded due to major data issues. In Part B, ppts who received Month 6 vaccination under protocol v6+ were randomized to mRNA-1273 or mRNA-1273.222. Ppts who received M6 vaccination before protocol v6 were not randomized because mRNA-1273.222 was unavailable.
Groups:
- Part A (Open-label): Study Group 1: Baseline HIV positive, baseline SARS-CoV-2 anti-S negative
- Part A (Open Label): Study Group 2: Baseline HIV positive, baseline SARS-CoV-2 anti-S positive
- Part A (Open-label): Study Group 3: Baseline HIV negative, baseline SARS-CoV-2 anti-S negative
- Part A (Open-label): Study Group 4: Baseline HIV negative, baseline SARS-CoV-2 anti-S positive
- Part B (Blinded): mRNA-1273 at Month 6: Received monovalent booster at Month 6
- Part B (Blinded): mRNA-1273.222 at Month 6: Received bivalent booster at Month 6
Period: Part A (Open-label)
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4 | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Started | 3740 | 7941 | 648 | 1672 | 0 | 0
Full Analysis Set (FAS) (All participants who received at least 1 vaccination.) | 3740 | 7941 | 648 | 1672 | 0 | 0
Safety Set (SS) (A subset of participants in FAS with solicited and unsolicited AEs collected.) | 558 | 692 | 99 | 142 | 0 | 0
Immunogenicity Set (IS) (A subset of participants who were sampled for cellular and humoral immunogenicity assays.) | 68 | 80 | 67 | 78 | 0 | 0
Per-Protocol Set (PP) (Participants in FAS who received the intended number of pre-month 6 vaccination doses with no major protocol deviations.) | 3604 | 7832 | 617 | 1607 | 0 | 0
Completed (Completed Part A and continued to Part B.) | 3648 | 7819 | 624 | 1606 | 0 | 0
Not Completed | 92 | 122 | 24 | 66 | 0 | 0
Not completed — Lost to Follow-up | 21 | 39 | 8 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 35 | 30 | 14 | 17 | 0 | 0
Not completed — Death | 23 | 28 | 1 | 9 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Participant Unable to Adhere to Visit Schedule | 10 | 18 | 0 | 7 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 3 | 4 | 1 | 5 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Period: Part B (Blinded)
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4 | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Started (Continued to Part B and received a Month 6 vaccination.) | 0 | 0 | 0 | 0 | 11243 | 2012
Received Month 6 Vaccination Set (FM6) (Participants in FAS who received a Month 6 vaccination, regardless of in or outside the randomization scheme.) | 0 | 0 | 0 | 0 | 11243 | 2012
Randomized Month 6 Set (RM6) (Participants in FAS who received a Month 6 vaccination under the randomization scheme.) | 0 | 0 | 0 | 0 | 1976 | 2012
Safety Set (SS) (A subset of participants in FM6 with solicited and unsolicited AEs collected.) | 0 | 0 | 0 | 0 | 1323 | 89
Immunogenicity Set (IS) (A subset of participants in FM6 who were sampled for cellular and humoral immunogenicity assays.) | 0 | 0 | 0 | 0 | 252 | 26
Full Per-Protocol Set (FPP) (Participants in RM6 who received their Month 0, Month 1 (if applicable), and Month 6 vaccinations as assigned with no major protocol deviations.) | 0 | 0 | 0 | 0 | 1960 | 2002
Completed | 0 | 0 | 0 | 0 | 2086 | 1676
Not Completed | 0 | 0 | 0 | 0 | 9157 | 336
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 219 | 88
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 91 | 55
Not completed — Death | 0 | 0 | 0 | 0 | 63 | 19
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 6 | 1
Not completed — Participant Unable to Adhere to Visit Schedule | 0 | 0 | 0 | 0 | 54 | 21
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 8682 | 125
Not completed — Other | 0 | 0 | 0 | 0 | 41 | 27

BASELINE CHARACTERISTICS:
Population: Overall SARS-CoV-2 neg indicates all anti-Spike (anti-S), anti-Nucleocapsid (anti-N), and virus detection (NAAT) neg. Overall SARS-CoV-2 pos indicates one of anti-S, anti-N, or NAAT pos. Only anti-S is used to determine study groups (SG) in the Participant Flow table. Anti-S, anti-N, and NAAT are used to determine analysis groups (AG) for analyses. SG1 (anti-S neg) includes AG1 (overall neg) and AG2-2 (overall pos). SG3 (anti-S neg) includes AG3 (overall neg) and AG4-2 (overall pos).
Groups:
- Part A (Open-label): Study Group 1, Analysis Group 1 (AG1): Participants in Study Group 1 who are baseline HIV positive and overall SARS-CoV-2 status negative
- Part A (Open-label): Study Group 1, Analysis Group 2-2 (AG2-2): Participants in Study Group 1 who are baseline HIV positive and overall SARS-CoV-2 status positive
- Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1): Participants in Study Group 2 who are baseline HIV positive and overall SARS-CoV-2 status positive
- Part A (Open-label): Study Group 3, Analysis Group 3 (AG3): Participants in Study Group 3 who are baseline HIV negative and overall SARS-CoV-2 status negative
- Part A (Open-label): Study Group 3, Analysis Group 4-2 (AG4-2): Participants in Study Group 3 who are baseline HIV negative and overall SARS-CoV-2 status positive
- Part A (Open-label): Study Group 4, Analysis Group 4-1 (AG4-1): Participants in Study Group 4 who are baseline HIV negative and overall SARS-CoV-2 status positive
- Total: Total of all reporting groups
Arm/Group | Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) | Part A (Open-label): Study Group 1, Analysis Group 2-2 (AG2-2) | Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1) | Part A (Open-label): Study Group 3, Analysis Group 3 (AG3) | Part A (Open-label): Study Group 3, Analysis Group 4-2 (AG4-2) | Part A (Open-label): Study Group 4, Analysis Group 4-1 (AG4-1) | Total
Number analyzed (Participants) | 2476 | 1264 | 7941 | 391 | 257 | 1672 | 14001
Age, Continuous [Median (Full Range); unit: years] | 39 [18 to 76] | 40 [18 to 73] | 39 [18 to 79] | 34 [19 to 84] | 39 [18 to 82] | 34 [18 to 86] | 39 [18 to 86]
Age, Customized [Count of Participants; unit: Participants]
  <=40 years | 1388 | 681 | 4484 | 260 | 136 | 1099 | 8048
  > years | 1088 | 583 | 3457 | 131 | 121 | 573 | 5953
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1676 | 911 | 6407 | 100 | 108 | 909 | 10111
  Male | 800 | 353 | 1534 | 291 | 149 | 763 | 3890
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 2475 | 1264 | 7940 | 391 | 257 | 1672 | 13999
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2433 | 1248 | 7848 | 358 | 233 | 1574 | 13694
  White | 0 | 0 | 1 | 4 | 0 | 0 | 5
  More than one race | 43 | 15 | 91 | 29 | 23 | 96 | 297
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Eswatini | 53 | 19 | 130 | 1 | 0 | 6 | 209
  Malawi | 188 | 44 | 408 | 1 | 0 | 1 | 642
  Botswana | 22 | 20 | 30 | 13 | 7 | 27 | 119
  South Africa | 1530 | 808 | 5438 | 337 | 212 | 1463 | 9788
  Uganda | 191 | 93 | 796 | 17 | 16 | 71 | 1184
  Zambia | 257 | 179 | 584 | 7 | 14 | 74 | 1115
  Kenya | 235 | 101 | 555 | 15 | 8 | 30 | 944

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With a First Occurrence of CDC-defined COVID-19 Starting 1 Day After Month 0 Dose Until Month 6 Dose in FAS Cohort Between Analysis Group 1 (AG1) and Analysis Group 2-1 (AG2-1)
Description: The CDC-based COVID-19 endpoint is defined as the first occurrence of symptomatic NAAT-confirmed COVID-19 based on the following criteria: 1. At least ONE of the following systemic or respiratory symptoms: Fever (≥ 38C), chills, cough, shortness of breath and/or difficulty breathing, fatigue, muscle and/or body aches [not related to exercise], headache, new loss of taste/smell, sore throat, congestion, runny nose, nausea, vomiting, or diarrhea, AND 2. At least ONE (post-baseline) nasal swab (or respiratory sample, if hospitalized) positive for SARS-CoV-2 by NAAT. Because additional NAAT testing was performed at Month 1 for AG1 but not AG2-1, NAAT results at Month 1 were not considered. 3. The symptom date and NAAT positive date must be within 14 days of each other. The date of a COVID-19 endpoint according to the CDC-based definition is the earlier date of a symptom and the date of positive NAAT that satisfy the criteria stated above. The CDC criteria do not require adjudication.
Time Frame: 1 day after Month 1 dose until Month 6 dose
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) | Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1)
Number analyzed (Participants) | 2476 | 7941
Participants | 76 | 151
Statistical Analysis 1: Comparison: Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) vs Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1); Test type: Other; p < .001, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.44 to 0.77]

2. Primary Outcome: Part A: Number of Participants With a First Occurrence of COVE-defined COVID-19 Starting 1 Day After Month 0 Dose Until Month 6 Dose in FAS Cohort Between Analysis Group 1 (AG1) and Analysis Group 2-1 (AG2-1
Description: The COVE-based COVID-19 endpoint is defined as the first occurrence of adjudicated symptomatic NAAT-confirmed COVID-19 based on the following criteria (same as in the Moderna mRNA-1273 COVE trial): 1. At least TWO of the following systemic symptoms: Fever ≥ 38◦C), chills, myalgia, headache, sore throat, new loss of taste or smell, OR 2. At least ONE of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, OR clinical or radiographical evidence of pneumonia, AND 3. At least ONE (post-baseline) nasal swab (or respiratory sample, if hospitalized) positive for SARS-CoV-2 by NAAT. The date of a COVID-19 endpoint is the later date of a symptom and the date of positive NAAT. The COVE criteria require adjudication.
Time Frame: 1 day after Month 0 dose until Month 6 dose
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) | Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1)
Number analyzed (Participants) | 2476 | 7941
Participants | 30 | 40
Statistical Analysis 1: Comparison: Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) vs Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1); Test type: Other; p = 0.003, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.29 to 0.78]

3. Primary Outcome: Part A: Number of Participants With a First Occurrence of COVE-based Severe COVID-19 Starting 1 Day After Month 0 Dose Until Month 6 Dose in FAS Between Analysis Group 1 (AG1) and Analysis Group 2-1 (AG2-1)
Description: The COVE-based severe COVID-19 endpoint is defined as the first occurrence of a confirmed case of COVE-based COVID-19, plus any of the following: 1. Clinical signs indicative of severe systemic illness, Respiratory Rate ≥ 30 per minute, Heart Rate ≥ 125 beats per minute, SpO2 ≤ 93% on room air at sea level or PaO2/FIO2 less than 300 mm Hg, OR 2. Respiratory failure or Acute Respiratory Distress Syndrome (ARDS), (defined as needing high-flow oxygen, noninvasive or mechanical ventilation, or ECMO), evidence of shock (systolic blood pressure less than 90 mmHg, diastolic BP less than 60 mmHg or requiring vasopressors), OR 3. Significant acute renal, hepatic, or neurologic dysfunction, OR 4. Admission to an intensive care unit or death. The severe COVE criteria require adjudication.
Time Frame: 1 day after Month 0 dose until Month 6 dose
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) | Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1)
Number analyzed (Participants) | 2476 | 7941
Participants | 5 | 4
Statistical Analysis 1: Comparison: Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) vs Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1); Test type: Other; p = 0.056, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.07 to 1.04]

4. Primary Outcome: Part B: Number of Participants With a First Occurrence of CDC-based COVID-19 Starting 14 Days After Month 6 Dose Until End of Follow up in RM6 Cohort Between Month 6 Monovalent and Bivalent Boost Groups
Description: The CDC-based COVID-19 endpoint is defined as the first occurrence of symptomatic NAAT-confirmed COVID-19 based on the following criteria: 1. At least ONE of the following systemic or respiratory symptoms: Fever (≥ 38C), chills, cough, shortness of breath and/or difficulty breathing, fatigue, muscle and/or body aches [not related to exercise], headache, new loss of taste/smell, sore throat, congestion, runny nose, nausea, vomiting, or diarrhea, AND 2. At least ONE (post-baseline) nasal swab (or respiratory sample, if hospitalized) positive for SARS-CoV-2 by NAAT. 3. The symptom date and NAAT positive date must be within 14 days of each other. The date of a COVID-19 endpoint according to the CDC-based definition is the earlier date of a symptom and the date of positive NAAT that satisfy the criteria stated above. The CDC criteria do not require adjudication.
Time Frame: 14 days after Month 6 dose until end of follow up (up to 18 months)
Population: Participants in FAS who received a Month 6 vaccination under the randomization scheme (RM6 cohort).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 1976 | 2012
Participants | 151 | 142
Statistical Analysis 1: Comparison: Part B (Blinded): mRNA-1273 at Month 6 vs Part B (Blinded): mRNA-1273.222 at Month 6; Test type: Other; p = 0.449, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.73 to 1.15]

5. Primary Outcome: Part B: Number of Participants With a First Occurrence of COVE-based COVID-19 Starting 14 Days After Month 6 Dose Until End of Follow up in RM6 Cohort Between Month 6 Monovalent and Bivalent Boost Group
Description: as for outcome 2
Time Frame: 14 days after Month 6 dose until end of follow up (up to 18 months)
Population: Participants in FAS who received a Month 6 vaccination under the randomization scheme (RM6 cohort).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 1976 | 2012
Participants | 8 | 7
Statistical Analysis 1: Comparison: Part B (Blinded): mRNA-1273 at Month 6 vs Part B (Blinded): mRNA-1273.222 at Month 6; Test type: Other; p = 0.23, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 2.29, 95% CI 2-sided [0.59 to 8.87]

6. Primary Outcome: Part B: Number of Participants With a First Occurrence of COVE-based Severe COVID-19 Starting 14 Days After Month 6 Dose Until End of Follow up in RM6 Cohort Between Month 6 Monovalent and Bivalent Groups
Description: Statistical analyses were not performed because there are fewer than 7 severe COVE-based severe COVID-19 starting 14 days after Month 6 dose until end of follow up in RM6 cohort.
Time Frame: 14 days after Month 6 dose until end of follow up (up to 18 months)
Population: Participants in FAS who received a Month 6 vaccination under the randomization scheme (RM6 cohort).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 1976 | 2012
Participants | 1 | 0

7. Primary Outcome: Part A: Number of Participants With Solicited Adverse Events in the Safety Subset
Description: All solicited adverse events/reactogenicity symptoms are followed until resolution and graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, dated July 2017. Local reacto symptoms collected are: erythema/redness, induration/swelling, lymphadenopathy, and pain/tenderness. Systemic reacto symptoms collected are: arthralgia, chills, fever, headache, malaise/fatigue, myalgia, and nausea.
Time Frame: Up to 7 days following Month 0 vaccination (all Study Groups) and up to 7 days following Month 1 vaccination (Study Groups 1 and 3)
Population: Safety subset.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4
Number analyzed (Participants) | 558 | 692 | 99 | 142
Participants
  Any Reacto After Month 0 Vaccination: Grade 0 | 320 | 428 | 68 | 82
  Any Reacto After Month 0 Vaccination: Grade 1 | 158 | 167 | 19 | 37
  Any Reacto After Month 0 Vaccination: Grade 2 | 79 | 87 | 11 | 22
  Any Reacto After Month 0 Vaccination: Grade 3 | 1 | 9 | 1 | 1
  Any Reacto After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Any Reacto After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Any Reacto After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Any Reacto After Month 1 Vaccination: Grade 0 | 352 | 0 | 65 | 0
  Any Reacto After Month 1 Vaccination: Grade 1 | 126 | 0 | 21 | 0
  Any Reacto After Month 1 Vaccination: Grade 2 | 59 | 0 | 9 | 0
  Any Reacto After Month 1 Vaccination: Grade 3 | 5 | 0 | 2 | 0
  Any Reacto After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Any Reacto After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Erythema/Redness After Month 0 Vaccination: Grade 0 | 533 | 671 | 95 | 130
  Erythema/Redness After Month 0 Vaccination: Grade 1 | 18 | 14 | 3 | 9
  Erythema/Redness After Month 0 Vaccination: Grade 2 | 7 | 6 | 1 | 3
  Erythema/Redness After Month 0 Vaccination: Grade 3 | 0 | 0 | 0 | 0
  Erythema/Redness After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Erythema/Redness After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Induration/Swelling After Month 0 Vaccination: Grade 0 | 508 | 636 | 96 | 125
  Induration/Swelling After Month 0 Vaccination: Grade 1 | 27 | 37 | 1 | 9
  Induration/Swelling After Month 0 Vaccination: Grade 2 | 23 | 18 | 2 | 8
  Induration/Swelling After Month 0 Vaccination: Grade 3 | 0 | 0 | 0 | 0
  Induration/Swelling After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Induration/Swelling After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Lymphadenopathy After Month 0 Vaccination: Grade 0 | 517 | 657 | 93 | 132
  Lymphadenopathy After Month 0 Vaccination: Grade 1 | 33 | 23 | 4 | 6
  Lymphadenopathy After Month 0 Vaccination: Grade 2 | 7 | 11 | 1 | 4
  Lymphadenopathy After Month 0 Vaccination: Grade 3 | 1 | 0 | 1 | 0
  Lymphadenopathy After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Lymphadenopathy After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Pain/Tenderness After Month 0 Vaccination: Grade 0 | 389 | 518 | 79 | 96
  Pain/Tenderness After Month 0 Vaccination: Grade 1 | 144 | 135 | 15 | 32
  Pain/Tenderness After Month 0 Vaccination: Grade 2 | 24 | 36 | 4 | 14
  Pain/Tenderness After Month 0 Vaccination: Grade 3 | 1 | 2 | 1 | 0
  Pain/Tenderness After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Pain/Tenderness After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Erythema/Redness After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Erythema/Redness After Month 1 Vaccination: Grade 0 | 532 | 0 | 96 | 0
  Erythema/Redness After Month 1 Vaccination: Grade 1 | 3 | 0 | 1 | 0
  Erythema/Redness After Month 1 Vaccination: Grade 2 | 7 | 0 | 0 | 0
  Erythema/Redness After Month 1 Vaccination: Grade 3 | 0 | 0 | 0 | 0
  Erythema/Redness After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Erythema/Redness After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Induration/Swelling After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Induration/Swelling After Month 1 Vaccination: Grade 0 | 509 | 0 | 94 | 0
  Induration/Swelling After Month 1 Vaccination: Grade 1 | 22 | 0 | 1 | 0
  Induration/Swelling After Month 1 Vaccination: Grade 2 | 11 | 0 | 2 | 0
  Induration/Swelling After Month 1 Vaccination: Grade 3 | 0 | 0 | 0 | 0
  Induration/Swelling After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Induration/Swelling After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Lymphadenopathy After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Lymphadenopathy After Month 1 Vaccination: Grade 0 | 513 | 0 | 90 | 0
  Lymphadenopathy After Month 1 Vaccination: Grade 1 | 24 | 0 | 5 | 0
  Lymphadenopathy After Month 1 Vaccination: Grade 2 | 5 | 0 | 2 | 0
  Lymphadenopathy After Month 1 Vaccination: Grade 3 | 0 | 0 | 0 | 0
  Lymphadenopathy After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Lymphadenopathy After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Pain/Tenderness After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Pain/Tenderness After Month 1 Vaccination: Grade 0 | 403 | 0 | 74 | 0
  Pain/Tenderness After Month 1 Vaccination: Grade 1 | 115 | 0 | 19 | 0
  Pain/Tenderness After Month 1 Vaccination: Grade 2 | 24 | 0 | 4 | 0
  Pain/Tenderness After Month 1 Vaccination: Grade 3 | 0 | 0 | 0 | 0
  Pain/Tenderness After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Pain/Tenderness After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Arthralgia After Month 0 Vaccination: Grade 0 | 488 | 621 | 88 | 127
  Arthralgia After Month 0 Vaccination: Grade 1 | 48 | 45 | 7 | 8
  Arthralgia After Month 0 Vaccination: Grade 2 | 22 | 23 | 3 | 7
  Arthralgia After Month 0 Vaccination: Grade 3 | 0 | 2 | 1 | 0
  Arthralgia After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Arthralgia After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Chills After Month 0 Vaccination: Grade 0 | 511 | 639 | 90 | 134
  Chills After Month 0 Vaccination: Grade 1 | 37 | 36 | 5 | 7
  Chills After Month 0 Vaccination: Grade 2 | 10 | 15 | 4 | 1
  Chills After Month 0 Vaccination: Grade 3 | 0 | 1 | 0 | 0
  Chills After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Chills After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Fever After Month 0 Vaccination: Grade 0 | 540 | 660 | 97 | 140
  Fever After Month 0 Vaccination: Grade 1 | 11 | 19 | 1 | 2
  Fever After Month 0 Vaccination: Grade 2 | 7 | 10 | 1 | 0
  Fever After Month 0 Vaccination: Grade 3 | 0 | 2 | 0 | 0
  Fever After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Fever After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Headache After Month 0 Vaccination: Grade 0 | 435 | 557 | 85 | 106
  Headache After Month 0 Vaccination: Grade 1 | 96 | 104 | 11 | 29
  Headache After Month 0 Vaccination: Grade 2 | 26 | 28 | 3 | 7
  Headache After Month 0 Vaccination: Grade 3 | 1 | 2 | 0 | 0
  Headache After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Headache After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Malaise/Fatigue After Month 0 Vaccination: Grade 0 | 443 | 558 | 84 | 109
  Malaise/Fatigue After Month 0 Vaccination: Grade 1 | 86 | 91 | 9 | 27
  Malaise/Fatigue After Month 0 Vaccination: Grade 2 | 29 | 39 | 5 | 6
  Malaise/Fatigue After Month 0 Vaccination: Grade 3 | 0 | 3 | 1 | 0
  Malaise/Fatigue After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Malaise/Fatigue After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Myalgia After Month 0 Vaccination: Grade 0 | 469 | 606 | 86 | 118
  Myalgia After Month 0 Vaccination: Grade 1 | 64 | 60 | 7 | 18
  Myalgia After Month 0 Vaccination: Grade 2 | 25 | 22 | 5 | 5
  Myalgia After Month 0 Vaccination: Grade 3 | 0 | 3 | 1 | 1
  Myalgia After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Myalgia After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Nausea After Month 0 Vaccination: Grade 0 | 507 | 633 | 92 | 131
  Nausea After Month 0 Vaccination: Grade 1 | 36 | 38 | 6 | 9
  Nausea After Month 0 Vaccination: Grade 2 | 15 | 19 | 1 | 2
  Nausea After Month 0 Vaccination: Grade 3 | 0 | 1 | 0 | 0
  Nausea After Month 0 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Nausea After Month 0 Vaccination: Missing | 0 | 1 | 0 | 0
  Arthralgia After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Arthralgia After Month 1 Vaccination: Grade 0 | 482 | 0 | 85 | 0
  Arthralgia After Month 1 Vaccination: Grade 1 | 42 | 0 | 11 | 0
  Arthralgia After Month 1 Vaccination: Grade 2 | 17 | 0 | 1 | 0
  Arthralgia After Month 1 Vaccination: Grade 3 | 1 | 0 | 0 | 0
  Arthralgia After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Arthralgia After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Chills After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Chills After Month 1 Vaccination: Grade 0 | 494 | 0 | 89 | 0
  Chills After Month 1 Vaccination: Grade 1 | 35 | 0 | 6 | 0
  Chills After Month 1 Vaccination: Grade 2 | 11 | 0 | 2 | 0
  Chills After Month 1 Vaccination: Grade 3 | 2 | 0 | 0 | 0
  Chills After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Chills After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Fever After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Fever After Month 1 Vaccination: Grade 0 | 527 | 0 | 93 | 0
  Fever After Month 1 Vaccination: Grade 1 | 10 | 0 | 2 | 0
  Fever After Month 1 Vaccination: Grade 2 | 4 | 0 | 2 | 0
  Fever After Month 1 Vaccination: Grade 3 | 1 | 0 | 0 | 0
  Fever After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Fever After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Headache After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Headache After Month 1 Vaccination: Grade 0 | 433 | 0 | 79 | 0
  Headache After Month 1 Vaccination: Grade 1 | 85 | 0 | 15 | 0
  Headache After Month 1 Vaccination: Grade 2 | 21 | 0 | 2 | 0
  Headache After Month 1 Vaccination: Grade 3 | 3 | 0 | 1 | 0
  Headache After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Headache After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Malaise/Fatigue After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Malaise/Fatigue After Month 1 Vaccination: Grade 0 | 428 | 0 | 75 | 0
  Malaise/Fatigue After Month 1 Vaccination: Grade 1 | 80 | 0 | 15 | 0
  Malaise/Fatigue After Month 1 Vaccination: Grade 2 | 30 | 0 | 5 | 0
  Malaise/Fatigue After Month 1 Vaccination: Grade 3 | 4 | 0 | 2 | 0
  Malaise/Fatigue After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Malaise/Fatigue After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Myalgia After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Myalgia After Month 1 Vaccination: Grade 0 | 464 | 0 | 84 | 0
  Myalgia After Month 1 Vaccination: Grade 1 | 62 | 0 | 11 | 0
  Myalgia After Month 1 Vaccination: Grade 2 | 14 | 0 | 1 | 0
  Myalgia After Month 1 Vaccination: Grade 3 | 2 | 0 | 1 | 0
  Myalgia After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Myalgia After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0
  Nausea After Month 1 Vaccination: number analyzed (Participants) | 543 | 0 | 98 | 0
  Nausea After Month 1 Vaccination: Grade 0 | 501 | 0 | 87 | 0
  Nausea After Month 1 Vaccination: Grade 1 | 33 | 0 | 9 | 0
  Nausea After Month 1 Vaccination: Grade 2 | 7 | 0 | 1 | 0
  Nausea After Month 1 Vaccination: Grade 3 | 1 | 0 | 0 | 0
  Nausea After Month 1 Vaccination: Grade 4 | 0 | 0 | 0 | 0
  Nausea After Month 1 Vaccination: Missing | 1 | 0 | 1 | 0

8. Primary Outcome: Part B: Number of Participants With Solicited Adverse Events in the Safety Subset
Description: as for outcome 7
Time Frame: Up to 7 days following Month 6 vaccination
Population: Participants in the safety subset who received a Month 6 vaccination, regardless of in or outside the randomization scheme, and with solicited and unsolicited AEs collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 1323 | 89
Participants
  Any Reacto After Month 6 Vaccination: Grade 0 | 877 | 71
  Any Reacto After Month 6 Vaccination: Grade 1 | 290 | 9
  Any Reacto After Month 6 Vaccination: Grade 2 | 135 | 6
  Any Reacto After Month 6 Vaccination: Grade 3 | 17 | 0
  Any Reacto After Month 6 Vaccination: Grade 4 | 0 | 0
  Any Reacto After Month 6 Vaccination: Missing | 4 | 3
  Erythema/Redness After Month 6 Vaccination: Grade 0 | 1282 | 85
  Erythema/Redness After Month 6 Vaccination: Grade 1 | 28 | 1
  Erythema/Redness After Month 6 Vaccination: Grade 2 | 9 | 0
  Erythema/Redness After Month 6 Vaccination: Grade 3 | 0 | 0
  Erythema/Redness After Month 6 Vaccination: Grade 4 | 0 | 0
  Erythema/Redness After Month 6 Vaccination: Missing | 4 | 3
  Induration/Swelling After Month 6 Vaccination: Grade 0 | 1254 | 83
  Induration/Swelling After Month 6 Vaccination: Grade 1 | 50 | 2
  Induration/Swelling After Month 6 Vaccination: Grade 2 | 15 | 1
  Induration/Swelling After Month 6 Vaccination: Grade 3 | 0 | 0
  Induration/Swelling After Month 6 Vaccination: Grade 4 | 0 | 0
  Induration/Swelling After Month 6 Vaccination: Missing | 4 | 3
  Lymphadenopathy After Month 6 Vaccination: Grade 0 | 1235 | 84
  Lymphadenopathy After Month 6 Vaccination: Grade 1 | 59 | 2
  Lymphadenopathy After Month 6 Vaccination: Grade 2 | 23 | 0
  Lymphadenopathy After Month 6 Vaccination: Grade 3 | 2 | 0
  Lymphadenopathy After Month 6 Vaccination: Grade 4 | 0 | 0
  Lymphadenopathy After Month 6 Vaccination: Missing | 4 | 3
  Pain/Tenderness After Month 6 Vaccination: Grade 0 | 1010 | 76
  Pain/Tenderness After Month 6 Vaccination: Grade 1 | 244 | 7
  Pain/Tenderness After Month 6 Vaccination: Grade 2 | 56 | 3
  Pain/Tenderness After Month 6 Vaccination: Grade 3 | 9 | 0
  Pain/Tenderness After Month 6 Vaccination: Grade 4 | 0 | 0
  Pain/Tenderness After Month 6 Vaccination: Missing | 4 | 3
  Arthralgia After Month 6 Vaccination: Grade 0 | 1182 | 80
  Arthralgia After Month 6 Vaccination: Grade 1 | 90 | 2
  Arthralgia After Month 6 Vaccination: Grade 2 | 39 | 4
  Arthralgia After Month 6 Vaccination: Grade 3 | 8 | 0
  Arthralgia After Month 6 Vaccination: Grade 4 | 0 | 0
  Arthralgia After Month 6 Vaccination: Missing | 4 | 3
  Chills After Month 6 Vaccination: Grade 0 | 1208 | 82
  Chills After Month 6 Vaccination: Grade 1 | 74 | 2
  Chills After Month 6 Vaccination: Grade 2 | 29 | 2
  Chills After Month 6 Vaccination: Grade 3 | 8 | 0
  Chills After Month 6 Vaccination: Grade 4 | 0 | 0
  Chills After Month 6 Vaccination: Missing | 4 | 3
  Fever After Month 6 Vaccination: Grade 0 | 1282 | 86
  Fever After Month 6 Vaccination: Grade 1 | 26 | 0
  Fever After Month 6 Vaccination: Grade 2 | 8 | 0
  Fever After Month 6 Vaccination: Grade 3 | 3 | 0
  Fever After Month 6 Vaccination: Grade 4 | 0 | 0
  Fever After Month 6 Vaccination: Missing | 4 | 3
  Headache After Month 6 Vaccination: Grade 0 | 1043 | 74
  Headache After Month 6 Vaccination: Grade 1 | 213 | 9
  Headache After Month 6 Vaccination: Grade 2 | 57 | 3
  Headache After Month 6 Vaccination: Grade 3 | 6 | 0
  Headache After Month 6 Vaccination: Grade 4 | 0 | 0
  Headache After Month 6 Vaccination: Missing | 4 | 3
  Malaise/Fatigue After Month 6 Vaccination: Grade 0 | 1076 | 76
  Malaise/Fatigue After Month 6 Vaccination: Grade 1 | 164 | 7
  Malaise/Fatigue After Month 6 Vaccination: Grade 2 | 70 | 3
  Malaise/Fatigue After Month 6 Vaccination: Grade 3 | 9 | 0
  Malaise/Fatigue After Month 6 Vaccination: Grade 4 | 0 | 0
  Malaise/Fatigue After Month 6 Vaccination: Missing | 4 | 3
  Myalgia After Month 6 Vaccination: Grade 0 | 1136 | 79
  Myalgia After Month 6 Vaccination: Grade 1 | 124 | 5
  Myalgia After Month 6 Vaccination: Grade 2 | 52 | 2
  Myalgia After Month 6 Vaccination: Grade 3 | 7 | 0
  Myalgia After Month 6 Vaccination: Grade 4 | 0 | 0
  Myalgia After Month 6 Vaccination: Missing | 4 | 3
  Nausea After Month 6 Vaccination: Grade 0 | 1211 | 82
  Nausea After Month 6 Vaccination: Grade 1 | 77 | 2
  Nausea After Month 6 Vaccination: Grade 2 | 29 | 2
  Nausea After Month 6 Vaccination: Grade 3 | 2 | 0
  Nausea After Month 6 Vaccination: Grade 4 | 0 | 0
  Nausea After Month 6 Vaccination: Missing | 4 | 3

9. Primary Outcome: Part A: Number of Participants With Unsolicited Adverse Events in the Safety Subset
Description: All unsolicited AEs are graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
Time Frame: Up to 28 days following Month 0 vaccination (all Study Groups) and up to 28 days following Month 1 vaccination (Study Groups 1 and 3)
Population: Safety subset.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4
Number analyzed (Participants) | 558 | 692 | 99 | 142
Participants
  None | 506 | 668 | 91 | 134
  Mild | 16 | 7 | 1 | 2
  Moderate | 30 | 17 | 7 | 5
  Severe | 6 | 0 | 0 | 1

10. Primary Outcome: Part B: Number of Participants With Unsolicited Adverse Events in the Safety Subset
Description: as for outcome 9
Time Frame: Up to 28 days following Month 6 vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 1323 | 89
Participants
  None | 1290 | 87
  Mild | 9 | 0
  Moderate | 17 | 1
  Severe | 5 | 1
  Death | 2 | 0

11. Primary Outcome: Part A: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is any AE that results in any of the following outcomes: death, a life-threatening adverse event, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect, or is medically important.
Time Frame: Up to Month 6
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4
Number analyzed (Participants) | 3740 | 7941 | 648 | 1673
Participants | 84 | 126 | 5 | 32

12. Primary Outcome: Part B: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 11
Time Frame: Day of Month 6 vaccination up to Month 18
Population: Participants who received a Month 6 vaccination, regardless of in or outside the randomization scheme, and with solicited and unsolicited AEs collected (FM6 cohort).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 11243 | 2012
Participants | 212 | 45

13. Primary Outcome: Part A: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Adverse events of special interest (AESI) were described in Appendix L of the protocol. AESI for this protocol include but are not limited to potential immune-mediated diseases.
Time Frame: Up to Month 6
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4
Number analyzed (Participants) | 3740 | 7941 | 648 | 1673
Participants | 36 | 59 | 4 | 19

14. Primary Outcome: Part B: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: as for outcome 13
Time Frame: Day of Month 6 vaccination up to Month 18
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
Number analyzed (Participants) | 11243 | 2012
Participants | 111 | 27

15. Secondary Outcome: Part A: Number of Participants With First CDC-based COVID-19 Occurrence From 1 Day After Month 0 Dose to Month 6 Dose in FAS Cohort, Comparing Baseline SARS-CoV-2 Negative vs Positive, Regardless of HIV Status
Description: as for outcome 1
Time Frame: 1 day after Month 0 dose until Month 6 dose
Population: FAS. Participants who are baseline overall SARS-CoV-2 negative regardless of HIV status are comprised of Analysis Groups 1 and 3. Those who are baseline overall SARS-CoV-2 positive regardless of HIV status are comprised of Analysis Groups 2-1 and 4-1. Of note, overall SARS-CoV-2 status negative indicates all anti-Spike (anti-S), anti-Nucleocapsid (anti-N), and virus detection (NAAT) negative. Overall SARS-CoV-2 status positive indicates one of anti-S, anti-N, or NAAT positive.
Measure: Count of Participants; unit: Participants
Groups:
- Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3): Participants who are overall SARS-CoV-2 negative at baseline regardless of HIV status
- Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1): Participants who are overall SARS-CoV-2 positive at baseline regardless of HIV status
Arm/Group | Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3) | Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1)
Number analyzed (Participants) | 2867 | 9613
Participants | 86 | 179
Statistical Analysis 1: Comparison: Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3) vs Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1); Test type: Other; p < .001, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.43 to 0.73]

16. Secondary Outcome: Part A: Number of Participants With First COVE-based COVID-19 Occurrence From 1 Day After Month 0 Dose to Month 6 Dose in FAS Cohort, Comparing Baseline SARS-CoV-2 Negative vs Positive, Regardless of HIV Statu
Description: as for outcome 2
Time Frame: 1 day after Month 0 dose until Month 6 dose
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3) | Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1)
Number analyzed (Participants) | 2867 | 9613
Participants | 34 | 45
Statistical Analysis 1: Comparison: Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3) vs Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1); Test type: Other; p < .001, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.27 to 0.68]

17. Secondary Outcome: Part A: Number of Participants With First COVE-based Severe COVID-19 Occurrence From 1 Day After Month 0 Dose to Month 6 Dose in FAS Cohort, Comparing Baseline SARS-CoV-2 Negative vs Positive, Regardless of HI
Description: as for outcome 3
Time Frame: 1 day after Month 0 dose until Month 6 dose
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3) | Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1)
Number analyzed (Participants) | 2867 | 9613
Participants | 7 | 6
Statistical Analysis 1: Comparison: Part A (Open-label): Analysis Group 1 (AG1) + Analysis Group 3 (AG3) vs Part A (Open-label): Analysis Group 2-1 (AG2-1) + Analysis Group 4-1 (AG4-1); Test type: Other; p = 0.02, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.09 to 0.82]

18. Secondary Outcome: Part B: Number of Participants With a First Occurrence of CDC-based COVID-19 Starting 14 Days After Month 6 Dose Until End of Follow up in RM6 Cohort Who Have Month 6 Hybrid Immunity Between Month 6 Monovalent and Bivalent Boost Groups
Description: The CDC-based COVID-19 endpoint is defined as the first occurrence of symptomatic NAAT-confirmed COVID-19 based on these criteria: 1. At least ONE of the following systemic or respiratory symptoms: Fever (≥ 38C), chills, cough, shortness of breath and/or difficulty breathing, fatigue, muscle and/or body aches [not related to exercise], headache, new loss of taste/smell, sore throat, congestion, runny nose, nausea, vomiting, or diarrhea, AND 2. At least ONE (post-baseline) nasal swab (or respiratory sample, if hospitalized) positive for SARS-CoV-2 by NAAT. 3. The symptom date and NAAT positive date must be within 14 days of each other. The date of a COVID-19 endpoint according to the CDC-based definition is the earlier date of a symptom and date of positive NAAT that satisfy the criteria stated above. The CDC criteria do not require adjudication.
Time Frame: 14 days after Month 6 dose until end of follow up (up to 18 months)
Population: Participants in FAS who received a Month 6 vaccination under the randomization scheme (RM6 cohort) and have Month 6 hybrid immunity. Hybrid immunity is defined as any evidence of prior SARS-CoV-2 infection up to the Month 6 visit, defined by meeting any of the following criteria: 1) baseline overall SARS-CoV-2 status positive, 2) at least one NAAT result at or prior to Month 6 is positive, or 3) at least one anti-NP tests at or prior to Month 6 is positive.
Measure: Count of Participants; unit: Participants
Groups:
- Part B (Blinded): Monovalent, Month 6 Hybrid Immunity: Participants who received mRNA1273 and have hybrid immunity at Month 6. Hybrid immunity is defined as any evidence of prior SARS-CoV-2 infection up to the Month 6 visit, defined by meeting any of the following criteria: 1) baseline overall SARS-CoV-2 status positive, 2) at least one NAAT result at or prior to Month 6 is positive, or 3) at least one anti-NP tests at or prior to Month 6 is positive.
- Part B (Blinded): Bivalent, Month 6 Hybrid Immunity: Participants who received mRNA1273.222 and have hybrid immunity at Month 6. Hybrid immunity is defined as any evidence of prior SARS-CoV-2 infection up to the Month 6 visit, defined by meeting any of the following criteria: 1) baseline overall SARS-CoV-2 status positive, 2) at least one NAAT result at or prior to Month 6 is positive, or 3) at least one anti-NP tests at or prior to Month 6 is positive.
Arm/Group | Part B (Blinded): Monovalent, Month 6 Hybrid Immunity | Part B (Blinded): Bivalent, Month 6 Hybrid Immunity
Number analyzed (Participants) | 1732 | 1759
Participants | 140 | 123
Statistical Analysis 1: Comparison: Part B (Blinded): Monovalent, Month 6 Hybrid Immunity vs Part B (Blinded): Bivalent, Month 6 Hybrid Immunity; Test type: Other; p = 0.218, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.67 to 1.09]

19. Secondary Outcome: Part B: Number of Participants With a First Occurrence of CDC-based COVID-19 Starting 14 Days After Month 6 Dose Until End of Follow up in RM6 Cohort Who Have Month 6 Vaccine Immunity Between Month 6 Monovalent and Bivalent Boost Group
Description: as for outcome 18
Time Frame: 14 days after Month 6 dose until end of follow up (up to 18 months)
Population: Participants in FAS who received a Month 6 vaccination under the randomization scheme (RM6 cohort) and have Month 6 vaccine immunity. Vaccine immunity is defined as absence of evidence of prior SARS-C
Measure: Count of Participants; unit: Participants
Groups:
- Part B (Blinded): Monovalent, Month 6 Vaccine Immunity: Participants who received mRNA1273 and have vaccine immunity at Month 6. Vaccine immunity is defined as absence of evidence of prior SARS-CoV-2 infection up to the Month 6 visit.
- Part B (Blinded): Bivalent, Month 6 Vaccine Immunity: Participants who received mRNA1273.222 and have vaccine immunity at Month 6. Vaccine immunity is defined as absence of evidence of prior SARS-CoV-2 infection up to the Month 6 visit.
Arm/Group | Part B (Blinded): Monovalent, Month 6 Vaccine Immunity | Part B (Blinded): Bivalent, Month 6 Vaccine Immunity
Number analyzed (Participants) | 244 | 253
Participants | 11 | 19
Statistical Analysis 1: Comparison: Part B (Blinded): Monovalent, Month 6 Vaccine Immunity vs Part B (Blinded): Bivalent, Month 6 Vaccine Immunity; Test type: Other; p = 0.135, Regression, Cox; Adjusted for variables expected to affect risk of future COVID-19 and evidence of prior SARS-CoV-2 exposure; Hazard Ratio (HR) = 1.78, 95% CI 2-sided [0.84 to 3.77]

20. Secondary Outcome: Part A: Geometric Mean Titers (GMTs) of SARS-CoV-2 Antibodies as Measured by Neutralizing Antibody (NAb) Assay
Description: Linear regression is used to provide covariate-adjusted point and 95% confidence interval estimation of geometric mean titers. Covariates adjusted are HIV status at baseline, age, sex at birth, and BMI.
Time Frame: Month 0, 4 weeks post final pre-Month 6 vaccination (peak timepoint)
Population: Per-protocol serum immunogenicity set with antibody marker data available at Month 0 and peak timepoint. Hybrid immunity is defined by one pre-Month 6 immunization after natural infection. Vaccine-induced immunity is defined by two pre-Month 6 immunizations for baseline overall SARS-CoV-2 negative ppts. The purpose is to summarize NAb responses by vaccine regimen (hybrid vs vaccine), as well as within people living with HIV (PWH) and people living without HIV (PWoH) respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/ml
Groups:
- Part A (Open-label): Hybrid Immunity: Baseline overall SARS-CoV-2 positive, 1 pre-Month 6 mRNA-1273 dose
- Part A (Open-label): Vaccine Immunity: Baseline overall SARS-CoV-2 negative, 2 mRNA-1273 pre-Month 6 doses
- Part A (Open-label): Hybrid Immunity, PWH: Baseline overall SARS-CoV-2 positive, 1 pre-Month 6 mRNA-1273 dose, baseline HIV positive
- Part A (Open-label): Hybrid Immunity, PWoH: Baseline overall SARS-CoV-2 positive, 1 pre-Month 6 mRNA-1273 dose, baseline HIV negative
- Part A (Open-label): Vaccine Immunity, PWH: Baseline overall SARS-CoV-2 negative, 2 mRNA-1273 pre-Month 6 doses, baseline HIV positive
- Part A (Open-label): Vaccine Immunity, PWoH: Baseline overall SARS-CoV-2 negative, 2 mRNA-1273 pre-Month 6 doses, baseline HIV negative
Arm/Group | Part A (Open-label): Hybrid Immunity | Part A (Open-label): Vaccine Immunity | Part A (Open-label): Hybrid Immunity, PWH | Part A (Open-label): Hybrid Immunity, PWoH | Part A (Open-label): Vaccine Immunity, PWH | Part A (Open-label): Vaccine Immunity, PWoH
Number analyzed (Participants) | 287 | 115 | 195 | 92 | 86 | 29
AU/ml
  Month 0 nAb-ID50 BA.4/5 | 348 [265 to 459] | 9 [7 to 12] | 324 [219 to 477] | 372 [227 to 583] | 9 [7 to 14] | 9 [6 to 15]
  Peak nAb-ID50 BA.4/5 | 4904 [3502 to 6846] | 705 [460 to 1065] | 5474 [3101 to 9417] | 4986 [2986 to 8350] | 996 [557 to 1726] | 326 [202 to 533]

21. Secondary Outcome: Part A: Geometric Mean Titers (GMTs) of SARS-CoV-2 Antibodies as Measured by Meso Scale Discovery-electrochemiluminescence Assay (MSD-ECL)
Description: as for outcome 20
Time Frame: Month 0, 4 weeks post final pre-Month 6 vaccination (peak timepoint)
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: AU/ml
Arm/Group | Part A (Open-label): Hybrid Immunity | Part A (Open-label): Vaccine Immunity | Part A (Open-label): Hybrid Immunity, PWH | Part A (Open-label): Hybrid Immunity, PWoH | Part A (Open-label): Vaccine Immunity, PWH | Part A (Open-label): Vaccine Immunity, PWoH
Number analyzed (Participants) | 287 | 115 | 195 | 92 | 86 | 29
AU/ml
  Month 0 IgG N Index | 52023 [38843 to 68767] | 5978 [4191 to 8489] | 52088 [33740 to 79760] | 48473 [33007 to 71126] | 4822 [3226 to 7397] | 5977 [4926 to 7573]
  Month 0 IgG Spike BA.5 | 17481 [13885 to 21634] | 480 [344 to 657] | 14893 [10481 to 21032] | 18066 [12261 to 25693] | 818 [546 to 1223] | 161 [129 to 196]
  Peak IgG Spike BA.5 | 205247 [178321 to 236883] | 126285 [102488 to 156924] | 188439 [159506 to 224439] | 232660 [170309 to 314805] | 130327 [99833 to 167232] | 77390 [65364 to 93101]

22. Secondary Outcome: Part A: Geometric Mean Titers of T-Cell Responses as Measured by Intracellular Cytokine Staining (ICS) Assay at Month 0
Description: as for outcome 20
Time Frame: Month 0
Population: Per-protocol PBMC immunogenicity set with cellular marker data available at Month 0. Hybrid immunity is defined by one pre-Month 6 immunization after natural infection. Vaccine-induced immunity is defined by two pre-Month 6 immunizations for baseline overall SARS-CoV-2 negative ppts. The purpose is to summarize NAb responses by vaccine regimen (hybrid vs vaccine), as well as within people living with HIV (PWH) and people living without HIV (PWoH) respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: % T-cells
Arm/Group | Part A (Open-label): Hybrid Immunity | Part A (Open-label): Vaccine Immunity | Part A (Open-label): Hybrid Immunity, PWH | Part A (Open-label): Hybrid Immunity, PWoH
Number analyzed (Participants) | 118 | 50 | 61 | 57
% T-cells
  Month 0 CD4+ IFNg/IL2 in response to BA.4-5 N | 0.0418 [0.0352 to 0.0505] | 0.0201 [0.0159 to 0.0257] | 0.0514 [0.0359 to 0.0762] | 0.035 [0.0283 to 0.0434]
  Month 0 CD4+ IFNg/IL2 in response to Spike BA.4/5 | 0.051 [0.0427 to 0.0601] | 0.0212 [0.0165 to 0.0272] | 0.0593 [0.0431 to 0.0804] | 0.0469 [0.0381 to 0.0573]
  Month 0 CD4+ IFNg/IL2/CD154 in response to BA.4-5 N | 0.0568 [0.0475 to 0.068] | 0.0256 [0.0194 to 0.0342] | 0.0671 [0.0464 to 0.0998] | 0.0491 [0.0398 to 0.0609]
  Month 0 CD4+ IFNg/IL2/CD154 in response to Spike BA.4/5 | 0.0757 [0.0638 to 0.0896] | 0.0298 [0.0226 to 0.039] | 0.0807 [0.0573 to 0.109] | 0.0737 [0.0595 to 0.0897]
  Month 0 CD8+ IFNg/IL2 in response to BA.4-5 N | 0.025 [0.0205 to 0.0307] | 0.0149 [0.0126 to 0.0183] | 0.0229 [0.0162 to 0.0333] | 0.0264 [0.0206 to 0.0347]
  Month 0 CD8+ IFNg/IL2 in response to Spike BA.4/5 | 0.0314 [0.0249 to 0.0401] | 0.0149 [0.0123 to 0.0183] | 0.0287 [0.0219 to 0.0384] | 0.0328 [0.0238 to 0.0459]

23. Secondary Outcome: Part A: Geometric Mean Titers of T-Cell Responses as Measured by Intracellular Cytokine Staining (ICS) Assay at Peak Timepoint
Description: as for outcome 20
Time Frame: 4 weeks post final pre-Month 6 vaccination (peak timepoint)
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: % T-cells
Arm/Group | Part A (Open-label): Hybrid Immunity | Part A (Open-label): Vaccine Immunity | Part A (Open-label): Hybrid Immunity, PWH | Part A (Open-label): Hybrid Immunity, PWoH | Part A (Open-label): Vaccine Immunity, PWH | Part A (Open-label): Vaccine Immunity, PWoH
Number analyzed (Participants) | 118 | 50 | 61 | 57 | 29 | 21
% T-cells
  Peak CD4+ IFNg/IL2 in response to BA.4-5 N | 0.0396 [0.0339 to 0.0468] | 0.0178 [0.0145 to 0.0223] | 0.0459 [0.034 to 0.0638] | 0.0354 [0.0293 to 0.0431] | 0.0269 [0.0178 to 0.0418] | 0.0135 [0.012 to 0.0156]
  Peak CD4+ IFNg/IL2 in response to Spike BA.4/5 | 0.2226 [0.1938 to 0.2531] | 0.2216 [0.1525 to 0.3053] | 0.2364 [0.1887 to 0.2925] | 0.214 [0.1766 to 0.2565] | 0.2463 [0.1331 to 0.4461] | 0.1704 [0.1539 to 0.1883]
  Peak CD4+ IFNg/IL2/CD154 in response to BA.4-5 N | 0.0548 [0.0465 to 0.0639] | 0.0242 [0.0186 to 0.0314] | 0.0588 [0.0433 to 0.0801] | 0.0513 [0.0416 to 0.0631] | 0.0362 [0.023 to 0.0585] | 0.0156 [0.0137 to 0.018]
  Peak CD4+ IFNg/IL2/CD154 in response to Spike BA.4/5 | 0.2786 [0.2454 to 0.3163] | 0.2883 [0.2077 to 0.3872] | 0.2943 [0.2404 to 0.3537] | 0.2681 [0.2217 to 0.3192] | 0.3138 [0.1734 to 0.5621] | 0.23 [0.2069 to 0.2551]
  Peak CD8+ IFNg/IL2 in response to BA.4-5 N | 0.024 [0.0197 to 0.0296] | 0.0148 [0.0127 to 0.0181] | 0.0222 [0.0158 to 0.0322] | 0.0254 [0.0199 to 0.0321] | 0.0138 [0.0116 to 0.0171] | 0.0157 [0.0142 to 0.0179]
  Peak CD8+ IFNg/IL2 in response to Spike BA.4/5 | 0.0481 [0.0381 to 0.061] | 0.0359 [0.0265 to 0.0478] | 0.0407 [0.0305 to 0.0552] | 0.0527 [0.0385 to 0.0733] | 0.0246 [0.0176 to 0.036] | 0.028 [0.021 to 0.0377]

24. Secondary Outcome: Part B: Geometric Mean Titers (GMTs) of SARS-CoV-2 Antibodies as Measured by Neutralizing Antibody Assay
Time Frame: Months 6 and 7
Population: Per-protocol serum immunogenicity set with antibody marker data available at Months 6 and 7. Hybrid immunity is defined by one pre-Month 6 immunization after natural infection. Vaccine-induced immunity is defined by two pre-Month 6 immunizations for baseline overall SARS-CoV-2 negative ppts.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/ml
Arm/Group | Part B (Blinded): Monovalent, Month 6 Hybrid Immunity | Part B (Blinded): Monovalent, Month 6 Vaccine Immunity | Part B (Blinded): Bivalent, Month 6 Hybrid Immunity | Part B (Blinded): Bivalent, Month 6 Vaccine Immunity
Number analyzed (Participants) | 74 | 26 | 75 | 25
AU/ml
  Month 6 ID50 Titer to BA.4/5: number analyzed (Participants) | 72 | 26 | 75 | 25
  Month 6 ID50 Titer to BA.4/5 | 750 [545.1 to 1031.9] | 1121.4 [603.5 to 2083.7] | 970.4 [709.8 to 1326.6] | 390.3 [189.6 to 803.5]
  Month 6 ID50 Titer to XBB.1.5: number analyzed (Participants) | 72 | 26 | 75 | 25
  Month 6 ID50 Titer to XBB.1.5 | 124.8 [86 to 181.1] | 169.2 [99.5 to 287.8] | 194 [127.9 to 294.3] | 80.1 [38.9 to 164.9]
  Month 6 ID80 Titer to BA.4/5: number analyzed (Participants) | 72 | 26 | 75 | 25
  Month 6 ID80 Titer to BA.4/5 | 127 [97.3 to 165.7] | 174.5 [93.9 to 324.2] | 150.4 [110 to 205.6] | 72.8 [38.7 to 136.9]
  Month 6 ID80 Titer to XBB.1.5: number analyzed (Participants) | 72 | 26 | 75 | 25
  Month 6 ID80 Titer to XBB.1.5 | 26.1 [19 to 35.9] | 34.4 [22.1 to 53.5] | 38.2 [26.5 to 55] | 21.9 [11.6 to 41.2]
  Month 7 ID50 Titer to BA.4/5: number analyzed (Participants) | 74 | 26 | 74 | 25
  Month 7 ID50 Titer to BA.4/5 | 2624.7 [2019.1 to 3411.9] | 2326.5 [1494.5 to 3621.6] | 4519.8 [3299.2 to 6191.9] | 1915.1 [849.9 to 4315.1]
  Month 7 ID50 Titer to XBB.1.5: number analyzed (Participants) | 74 | 26 | 74 | 25
  Month 7 ID50 Titer to XBB.1.5 | 542.4 [375.7 to 783.1] | 607.9 [327.2 to 1129.5] | 1521.5 [1000 to 2315] | 577.6 [234.2 to 1424.4]
  Month 7 ID80 Titer to BA.4/5: number analyzed (Participants) | 74 | 26 | 74 | 25
  Month 7 ID80 Titer to BA.4/5 | 546.9 [420.7 to 710.9] | 511.5 [300.8 to 869.9] | 1033.6 [754.5 to 1416] | 369.3 [179.4 to 760.3]
  Month 7 ID80 Titer to XBB.1.5: number analyzed (Participants) | 74 | 26 | 74 | 25
  Month 7 ID80 Titer to XBB.1.5 | 122.3 [84.7 to 176.6] | 126.8 [74.6 to 215.7] | 326.5 [214.6 to 496.8] | 115.5 [46.8 to 284.8]

25. Secondary Outcome: SARS-CoV-2 Viral Persistence and Evolution Among Participants Virologically Diagnosed With SARS-CoV-2
Description: Participants were considered to have persistent SARS-CoV-2 NAAT positivity if they had positive swabs lasting >= 50 days during a single infection. A single infection was assumed unless the participant had a positive NAAT following either a single negative NAAT by >= 90 days or two consecutive negative NAATs over any time interval, in which case it was considered a reinfection. In Part A, the first NAAT+ on or before the Month 6 dose for each ppt was considered. In Part B, the first NAAT+ after the Month 6 dose for each ppt was considered. Analysis of viral evolution was not done due to termination of resources for evaluation.
Time Frame: Participants testing positive for SARS-CoV-2 had additional nasab swabs taken fortnightly until testing negative, up to a maximum of 18 months
Population: Participants who are NAAT+ in the FAS cohort in part A. Participants who are NAAT+ in the RM6 cohort in part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part B (Blinded): HIV+ Monovalent: Participants who are baseline HIV positive and received mRNA1273 at Month 6
- Part B (Blinded): HIV+ Bivalent: Participants who are baseline HIV positive and received mRNA1273.222 at Month 6
- Part B (Blinded): HIV- Monovalent: Participants who are baseline HIV negative and received mRNA1273 at Month 6
- Part B (Blinded): HIV- Bivalent: Participants who are baseline HIV negative and received mRNA1273.222 at Month 6
Arm/Group | Part A (Open-label): Study Group 1, Analysis Group 1 (AG1) | Part A (Open-label): Study Group 1, Analysis Group 2-2 (AG2-2) | Part A (Open-label): Study Group 2, Analysis Group 2-1 (AG2-1) | Part A (Open-label): Study Group 3, Analysis Group 3 (AG3) | Part A (Open-label): Study Group 3, Analysis Group 4-2 (AG4-2) | Part A (Open-label): Study Group 4, Analysis Group 4-1 (AG4-1) | Part B (Blinded): HIV+ Monovalent | Part B (Blinded): HIV+ Bivalent | Part B (Blinded): HIV- Monovalent | Part B (Blinded): HIV- Bivalent
Number analyzed (Participants) | 220 | 333 | 597 | 27 | 52 | 132 | 229 | 200 | 55 | 46
percentage of participants | 2.27 [0.97 to 5.21] | 3.3 [1.85 to 5.82] | 1.17 [0.57 to 2.40] | 0 [0.00 to 12.46] | 3.85 [1.06 to 12.98] | 0.76 [0.13 to 4.17] | 1.31 [0.45 to 3.78] | 0 [0.00 to 1.88] | 0 [0.00 to 6.53] | 0 [0.00 to 7.71]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected for 7 days following each vaccination. Unsolicited AEs were collected for 28 days following each vaccination. Serious AEs were collected until end of follow up (up to 18 months).
Description: All cause mortality and serious AEs were collected and reported on all participants in the FAS cohort. Other AEs were collected and reported on safety subset participants in the FAS cohort for Part A and on safety subset participants in the FM6 cohort for Part B. In each AE table, AEs following Month 0 and/or Month 1 vaccination were reported for Part A and AEs following Month 6 vaccination were reported for Part B.
Arm/Group | Part A (Open-label): Study Group 1 | Part A (Open Label): Study Group 2 | Part A (Open-label): Study Group 3 | Part A (Open-label): Study Group 4 | Part B (Blinded): mRNA-1273 at Month 6 | Part B (Blinded): mRNA-1273.222 at Month 6
All-Cause Mortality (participants affected / at risk) | 24/3740 | 31/7941 | 1/648 | 9/1672 | 63/11243 | 19/2012
Serious Adverse Events (participants affected / at risk) | 84/3740 | 126/7941 | 5/648 | 32/1672 | 212/11243 | 45/2012
Other Adverse Events (participants affected / at risk) | 308/558 | 270/692 | 47/99 | 62/142 | 450/1323 | 15/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Open-label): Study Group 1 (N=3740) | Part A (Open Label): Study Group 2 (N=7941) | Part A (Open-label): Study Group 3 (N=648) | Part A (Open-label): Study Group 4 (N=1672) | Part B (Blinded): mRNA-1273 at Month 6 (N=11243) | Part B (Blinded): mRNA-1273.222 at Month 6 (N=2012)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fanconi syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 13 (13) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Type IV hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complicated malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis AIDS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapulmonary Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Eye infection syphilitic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 1 (1)
HIV peripheral neuropathy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIV wasting syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIV-associated neurocognitive disorder (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Male genital tract tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis meningococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Meningoencephalitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (9) | 6 (6) | 0 (0) | 3 (3) | 13 (13) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 12 (12) | 0 (0) | 1 (1) | 8 (8) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Uterine rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain stem syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Abortion spontaneous complicated (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Factitious disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (Open-label): Study Group 1 (N=558) | Part A (Open Label): Study Group 2 (N=692) | Part A (Open-label): Study Group 3 (N=99) | Part A (Open-label): Study Group 4 (N=142) | Part B (Blinded): mRNA-1273 at Month 6 (N=1323) | Part B (Blinded): mRNA-1273.222 at Month 6 (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Solicited) (Blood and lymphatic system disorders) | 64 (70) | 34 (34) | 9 (13) | 10 (10) | 84 (84) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid rash (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Solicited) (Gastrointestinal disorders) | 82 (92) | 58 (58) | 13 (17) | 11 (11) | 108 (108) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (Solicited) (General disorders) | 82 (95) | 52 (52) | 12 (17) | 8 (8) | 111 (111) | 4 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (Solicited) (General disorders) | 178 (229) | 133 (133) | 27 (37) | 33 (33) | 243 (243) | 10 (10)
Influenza like illness (General disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (Solicited) (General disorders) | 221 (308) | 173 (173) | 34 (43) | 46 (46) | 309 (309) | 10 (10)
Swelling (Solicited) (General disorders) | 72 (83) | 55 (55) | 4 (6) | 17 (17) | 65 (65) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea faciei (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Solicited) (Investigations) | 30 (33) | 31 (31) | 5 (6) | 2 (2) | 37 (37) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 112 (130) | 70 (70) | 17 (23) | 15 (15) | 137 (137) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 130 (167) | 85 (85) | 18 (26) | 24 (24) | 183 (183) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Headache (Solicited) (Nervous system disorders) | 182 (232) | 134 (134) | 25 (32) | 36 (36) | 276 (276) | 12 (12)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Solicited) (Skin and subcutaneous tissue disorders) | 33 (35) | 20 (20) | 5 (5) | 12 (12) | 37 (37) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Informed Consent Form (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT05168813/Prot_ICF_000.pdf
  • Statistical Analysis Plan: Pre-Month 6 Efficacy SAP (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT05168813/SAP_001.pdf
  • Statistical Analysis Plan: Post-Month 6 Efficacy SAP (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT05168813/SAP_002.pdf